CLINICAL TRIAL: NCT06615050
Title: A Randomized, Multicenter, Phase III Trial of Tacrolimus/Methotrexate/Ruxolitinib Versus Post-Transplant Cyclophosphamide/Tacrolimus/Mycophenolate Mofetil in Non-Myeloablative/Reduced Intensity Conditioning Allogeneic Peripheral Blood Stem Cell Transplantation
Brief Title: A Study of Tacrolimus/Methotrexate/Ruxolitinib Versus Post-Transplant Cyclophosphamide/Tacrolimus/Mycophenolate Mofetil in Non-Myeloablative/Reduced Intensity Conditioning Allogeneic Peripheral Blood Stem Cell Transplantation (BMT CTN 2203)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB18424-370; BMT CTN Protocol 2203 (Other: Blood and Marrow Transplant Clinical Trials Network)
Record Dates: First submitted 2024-09-06; First posted 2024-09-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: Graft-versus-host Disease (GVHD); Chronic GvHD (cGvHD); steroid-refractory; ruxolitinib; Janus kinase inhibitor
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Tacrolimus; Triamcinolone; Methotrexate; ruxolitinib; Cyclophosphamide; Mycophenolic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dose Finding Run-In Group 1: Tac/MTX/Ruxolitnib Dose 1 (Experimental): Tacrolimus/ methotrexate/ ruxolitinib (Tac/MTX/Rux) at the protocol defined doses.
  Interventions: Drug: Tacrolimus (Tac); Drug: Methotrexate (MTX); Drug: Ruxolitinib (Rux)
- Dose Finding Run-In Group 2: Tac/MTX/Ruxolitnib Dose 2 (Experimental): Tacrolimus/ methotrexate/ ruxolitinib (Tac/MTX/Rux) at the protocol defined doses.
  Interventions: Drug: Tacrolimus (Tac); Drug: Methotrexate (MTX); Drug: Ruxolitinib (Rux)
- Main Study Group A: Tac/MTX/Ruxolitnib (Experimental): Tacrolimus/ methotrexate/ ruxolitinib (Tac/MTX/Rux) at the protocol defined doses.
  Interventions: Drug: Tacrolimus (Tac); Drug: Methotrexate (MTX); Drug: Ruxolitinib (Rux)
- Main Study Group B: PTCy/Tac/MMF (Active Comparator): Post-transplant cyclophosphamide/ tacrolimus/ mycophenolate mofetil (PTCy/Tac/MMF) at the protocol defined doses.
  Interventions: Drug: Tacrolimus (Tac); Drug: Cyclophosphamide; Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Tacrolimus (Tac) — Tablet or intravenously (IV)
Drug: Methotrexate (MTX) — Intravenously (IV)
  Arms: Dose Finding Run-In Group 1: Tac/MTX/Ruxolitnib Dose 1; Dose Finding Run-In Group 2: Tac/MTX/Ruxolitnib Dose 2; Main Study Group A: Tac/MTX/Ruxolitnib
Drug: Ruxolitinib (Rux) — Tablet
  Other Names: Jakafi, INCB018424
  Arms: Dose Finding Run-In Group 1: Tac/MTX/Ruxolitnib Dose 1; Dose Finding Run-In Group 2: Tac/MTX/Ruxolitnib Dose 2; Main Study Group A: Tac/MTX/Ruxolitnib
Drug: Cyclophosphamide — Intravenously (IV)
  Arms: Main Study Group B: PTCy/Tac/MMF
Drug: Mycophenolate mofetil (MMF) — Tablet or intravenously (IV)
  Arms: Main Study Group B: PTCy/Tac/MMF

SUMMARY:
The purpose of this study is to assess Tacrolimus/Methotrexate/Ruxolitinib versus Post-Transplant Cyclophosphamide/Tacrolimus/Mycophenolate Mofetil in Non-Myeloablative/Reduced Intensity Conditioning Allogeneic Peripheral Blood Stem Cell Transplantation

ELIGIBILITY:
Inclusion Criteria:

* Age 18.0 years or older at the time of enrollment.
* Participants undergoing allogeneic HCT for one of the following indications:

  * Acute leukemia or chronic myelogenous leukemia with no circulating blasts and with less than 5% blasts in the bone marrow. Therapy related myeloid neoplasms are allowed.
  * Myelodysplasia/chronic myelomonocytic leukemia with no circulating blasts and with less than 10% blasts in the bone marrow (higher blast percentage allowed in MDS due to lack of differences in outcomes with < 5% versus 5-10% blasts in this disease). Therapy related myeloid neoplasms are allowed.
  * Lymphoma [follicular lymphoma, Hodgkin lymphoma, diffuse large B cell lymphoma, mantle cell lymphoma, peripheral T-cell lymphoma, angioimmunoblastic T-cell lymphoma and anaplastic large cell lymphoma].
* Planned NMA/reduced intensity conditioning regimen.
* Participants must have a related or unrelated PBSC donor as follows:

  * Sibling donor must be a 6/6 match for HLA-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing and must be willing to donate peripheral blood stem cells and meet institutional criteria for donation. HLA-matched parents and children may be used as donors.
  * Unrelated donor must be a 7/8 or 8/8 match at HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing. Unrelated donor must be willing to donate peripheral blood stem cells and meet NMDP criteria for donation.
  * Donor selection must comply with 21 CFR 1271.
* Cardiac function: Left ventricular ejection fraction at least 45%.
* Estimated creatinine clearance greater than 60 ml/min using the 2021 CKD-EPI formula or 24-hour urine creatinine clearance.
* Pulmonary function: DLCO corrected for hemoglobin at least 40% and FEV1 predicted at least 50%.
* Liver function: AST/ALT < 3x ULN; Total bilirubin < 2 mg/dL excluding Gilbert's syndrome or hemolysis.
* Karnofsky Performance Score of at least 60%.
* Female participants (unless postmenopausal for at least one year before the screening visit, or surgically sterilized), agree to practice two effective methods of contraception at the same time, or agree to completely abstain from heterosexual intercourse, from the time of signing the informed consent through 15 months post-transplant. Fertility preservation methods will be left to institutional standards.
* Male participants (even if surgically sterilized), of partners of women of childbearing potential must agree to one of the following: practice effective barrier contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 15 months post-transplant.
* Plans for the use of targeted small molecule inhibitor post-transplant maintenance therapy must be disclosed upon enrollment and must be used irrespective of the outcome of the randomization. Planned use of investigational maintenance agents is not permitted. Planned hypomethylating agents as maintenance therapy is not permitted.
* Voluntary written consent obtained prior to the performance of any study-related procedure that is not a part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.

Exclusion Criteria:

* Prior allogeneic transplant.
* Active CNS involvement by malignant cells.
* Participants with secondary AML arising from myeloproliferative neoplasms or overlap syndromes, including CMML and MDS/MPN syndromes; participants with secondary AML arising from myelodysplastic neoplasm are eligible.
* Participants with primary myelofibrosis.
* Participants with uncontrolled bacterial, viral, or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
* Active or inadequately treated latent infection with Mycobacterium tuberculosis (i.e., TB).
* Presence of clinically significant fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated.
* Participants seropositive for human immunodeficiency virus (HIV) with detectable viral load. HIV+ participants with an undetectable viral load on antiviral therapy are eligible.
* Evidence of uncontrolled hepatitis B virus (HBV) or hepatitis C virus (HCV). The study allows:

  * Positive HBV serology with undetectable viral load and ongoing antiviral prophylaxis to prevent potential HBV reactivation.
  * Positive HCV serology with quantitative PCR for plasma HCV RNA below the lower limit of detection, with or without concurrent antiviral HCV treatment.
* Arterial or venous thrombosis including DVT, PE, stroke, and myocardial infarction within six (6) months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia. Catheter-associated DVT is not exclusionary.
* Female participants who are pregnant (as per institutional practice) or lactating.
* Participants with a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Participants with prior malignancies except resected non-melanoma skin cancer or treated cervical carcinoma in situ. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously must be reviewed and approved by the Protocol Officer or Chairs.
* Planned use of ATG or alemtuzumab in conditioning regimen.
* Planned use of prophylactic donor leukocyte infusions.
* Prior use of ruxolitinib.
* Prior use of immune checkpoint inhibitors (i.e., PD1, PDL1, CTLA4 modulators) within six (6) months prior to conditioning.
* For participants with 7/8 HLA-matched donors:

  * Donor specific antibodies (DSAs) directed at the mismatched donor allele.
  * Any use of desensitization protocols.
* Treatment with any other Investigational Medicinal Product (IMP) is not allowed while on study treatment. An IMP is defined as medications without any known FDA or EMA approved indications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2031-01-17 (Estimated); Study Completion 2031-01-17 (Estimated)

PRIMARY OUTCOMES:
GVHD-free survival (GFS) | Up to 24 months post-transplant (Day 0)
  GFS will be defined as the elapsed time between the date of transplant to Grade III-IV acute graft-versus host disease (GVHD), chronic GVHD requiring systemic immune suppression, or death by any cause.

SECONDARY OUTCOMES:
GVHD/relapse or Progression-free Survival (GRFS) | Up to 24 months post-transplant (Day 0)
  Defined as Grade III-IV acute GVHD, chronic GVHD requiring systemic immune suppression, underlying disease relapse or progression, or death by any cause.
Incidence of chronic GVHD | Up to 24 months post-transplant (Day 0)
  Defined by the protocol.
Incidence of acute grade 2-4 and 3-4 graft versus host disease (GVHD) | Up to 24 months post-transplant (Day 0)
  Defined by the protocol.
Time to neutrophil and platelet recovery | Up to 24 months post-transplant (Day 0)
  Defined by the Protocol.
Donor Cell Engraftment | Up to 24 months post-transplant (Day 0)
  Defined by the protocol.
Cumulative incidence of primary and secondary graft failure | Day 28 and up to 2 years post-transplant (Day 0)
  Primary graft failure is defined as no neutrophil recovery to > 500 cells/μL by Day 28 post HSCT. Secondary graft failure is defined as initial neutrophil engraftment followed by subsequent decline in absolute neutrophil counts < 500 cells/μL, unresponsive to growth factor therapy, but cannot be explained by disease relapse or medications up to two years post-transplant.
Disease Relapse or Progression | Up to 24 months post-transplant (Day 0)
  Defined by the protocol.
Non-relapse Mortality | Up to 24 months post-transplant (Day 0)
  Defined as death without evidence of disease progression or recurrence.
Toxicity and Infections | Up to 24 months post-transplant (Day 0)
  All Grade 2-5 toxicities according to CTCAE, version 5.0 will be tabulated for each intervention arm. The proportion of participants developing at least a Grade 2 or higher toxicity across intervention arms will be compared.
Disease-Free Survival | Up to 24 months post-transplant (Day 0)
  Defined as the time from date of transplant to death or relapse/progression, whichever comes first.
Overall Survival | Up to 24 months post-transplant (Day 0)
  Defined as the time interval between date of transplant and death from any cause.
Modified Lee Chronic GVHD Symptom Scale (mLSS) | Up to 24 months post-transplant (Day 0)
  The modified Lee chronic GVHD symptom scale (mLSS) is a 28 item measure with seven domains referent to the past seven days: skin, mouth, eye, lung, psychoemotional, vitality and nutrition.
Individual Symptom Scale: Modified Medical Research Council (mMRC) Dyspnea scale | Up to 24 months post-transplant (Day 0)
  mMRC dyspnea scale assesses the degree of functional disability due to dyspnea.
Individual Symptom Scale: Two items from a protocol defined survey | Up to 24 months post-transplant (Day 0)
  Two items from a protocol defined survey are used to measure hemorrhagic cystitis symptom burden.
Individual Symptom Scale: Oral Health Impact Profile (OHIP) | Up to 24 months post-transplant (Day 0)
  OHIP measures dysfunction, discomfort and disability caused by oral conditions.
Individual Symptom Scale: Ocular Surface Disease Index (OSDI) | Up to 24 months post-transplant (Day 0)
  OSDI measures symptoms and vision effects of dry eye disease.
Work Productivity and Impairment Questionnaire (WPAI) | Up to 24 months post-transplant (Day 0)
  WPAI measures the impact on ability to work and perform regular activities.
Comprehensive Score for Financial Toxicity (COST) | Up to 24 months post-transplant (Day 0)
  COST measures the impacts of treatment on finances and economic status of the patient households.
Patient-Reported Economic, Income and Insurance Data (PREIID) | Up to 24 months post-transplant (Day 0)
  PREIID measures the impacts of treatment on finances and economic status of the patient households.
Patient Reported Caregiver Assessment (PRCA) | Up to 24 months post-transplant (Day 0)
  PRCA measures the type of support provided by caregivers, and the economic burden to patient caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (28):
- United States (28):
  - Stanford Cancer Center, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital Authority, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, North Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study of Tacrolimus/Methotrexate/Ruxolitinib Versus Post-Transplant Cyclophosphamide/Tacrolimus/Mycophenolate Mofetil in Non-Myeloablative/Reduced Intensity Conditioning Allogeneic Peripheral Blood Stem Cell Transplantation (BMT CTN 2203) — https://incyteclinicaltrials.com/studies/incb18424-370